CLINICAL TRIAL: NCT03601481
Title: Mise en Place et Validation d'un Logiciel de Télémédecine Permettant l'Automatisation du Traitement Des Examens IRM Des Infarctus du Myocarde en Phase Aigue
Brief Title: Implementation and Validation of Telemedicine Software for the Automation of MRI Examinations of Acute Myocardial Infarctions
Acronym: TELECARD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2012/36
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myocardial Infarction
Keywords: telemedicine; cardiac images
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validation of a telemedicine software application for an automated treatment of cardio-vascular MRI completely identical for both CHUs.

Providing the software application to other CHU seeking a tool suitable for multi-centric studies.

DETAILED DESCRIPTION:
1. Scientific context:

   Cardiac MRI has become a standard technique for determining the size of myocardial infarction as well as evaluating myocardial function and perfusion. However, the quantitative analysis of the images targeted on the left and right ventricles relies on computer treatments often manual so tedious and dependent on the user, or at best semi-automatic. The absence of a completely automated method limits the extraction of quantitative and reproducible parameters for each patient, which is necessary for the follow-up of patients who have had an acute myocardial infarction.
2. Objective (s):

   The goal is to integrate in a telemedicine software solution (partnership with the company Covalia) an automated method of processing these data completely identical for both CHUs. This development could be made available to other UHC seeking a tool suitable for multicenter studies.
3. Materials and Methods:

An engineer will be recruited to develop algorithms for robust, reliable and ergonomic software for the study of myocardial function and perfusion. The software will be accessible by users via the internet, and will integrate all the security and personal protection constraints that a telemedicine tool requires. The telemedicine aspect will be done in partnership with the company Covalia, which obtained for its software solutions CE marking thanks to an organization ISO 13485 applied to the whole of the company.

The images used for the realization of the software will be taken from the Besançon patient examinations included in the previous PHRC (1) and will be used after anonymisation.

Validation of the software will be based on current BioCard PHRC examinations in Dijon and Besançon. This study concerning the implementation and the validation of a software, a hundred of cases will be included in order to obtain a sufficient representation of the included population (ie sufficient observable variability) to validate the technical characteristics of the software (reliability, reproducibility, sensitivity, precision).

The software will automatically provide the calculation of tele-diastolic and tele-systolic volumes, ejection fraction, thickness and myocardial thickening. In addition, the study of myocardial infusion after injection of a contrast medium will consist of the construction of parametric perfusion maps, as well as an automatic determination of myocardial viability. The development of the computer tool will be based on the software "Quantified Imaging Resource", developed by Alain Lalande and Alexandre Comte and whose results have already been the subject of publications.

The aforementioned parameters will be calculated automatically (with the software) and manually (2 experts will perform these calculations). The results will then be compared and analyzed by the statisticians of the Besançon and Dijon clinical investigation centers

(1) : Détermination du taux et du type de progéniteurs vasculaires dans l'infarctus myocardique avec et sans sus décalage du segment ST - 2005 - Dr Meneveau (cardiologie)

4- Expected results and perspectives (less than 30 words)

* Complete software development and validation on the BioCard PHRC exams.
* Integration of the software in a tele-medicine application.
* Submission of at least two articles for international journals.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 75 yeras
* heart attack with medical treatment within 12 hours
* heart attack with or without segment S-T gap

Exclusion Criteria:

* cardiogenic choc
* medical history with heart attack,
* medical history with left ventricle dysfonction (ejection fraction< 45%),
* medical history with clinic manifestations of heart failure,
* medical history with surgical coronary revascularisation in the last 6 months,
* congenital cardiopathy, myocardiopathy,
* evolutive infection syndrome (HIV, VHB, VHC),
* chronic inflammatory pathology,
* leucopenia, thrombopenia, anemia,
* medical history with treatment by G-CSF; EPO; GM-CSF,
* stasis trouble, evolutive hemorragic syndrome, transfusion,
* renal insuffisance (clearance MDRD < 60ml/min),
* renal insuffisance with creatinin > 120 µmol/L,
* hepatic insuffisance,
* medical history of cancer or pathology with life expectancy < 1 year,
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient with heart attack
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Precision of the localisation of endocardic and epicardic edge | Day 2
  Validation of a software telemedecine for automatic treatment of cardio-vascular MRI
Volume of myocardic cavity | Day 2
Ejection fraction | Day 2
Weight of the myocard | Day 2
Thickness of the myocard | Day 2
Precision of the localisation of endocardic and epicardic edge | 6 months
Volume of myocardic cavity | 6 months
Weight of the myocard | 6 months
Thickness of the myocard | 6 months